CLINICAL TRIAL: NCT05915975
Title: Integrated Behavioral Healthcare for Low-Income Ethnic Minority Youth With Type 1 Diabetes
Brief Title: Integrated Behavioral Healthcare for Youth With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Luiza Vianna Mali, Assistant Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20230308
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Care Coordinated with Medical Care (Experimental): Participants in this group will work with a study team member for four months to improve your skills to manage diabetes, to strengthen the child-caregiver relationship, and/or to address emotional challenges that your child might be experiencing.
  Interventions: Behavioral: Behavioral Care Coordinated with Medical Care Intervention
- Behavioral Care Not Coordinated with Medical Care (Active Comparator): Participants will receive the standard of care treatment for four months plus a list of clinics that accept their insurance.
  Interventions: Behavioral: Behavioral Care Not Coordinated with Medical Care Intervention

INTERVENTIONS:
Behavioral: Behavioral Care Coordinated with Medical Care Intervention — Participants will be meeting with a behavioral health provider during their clinic visit. Subsequent visits can be held either via telehealth or in-person. Participants should expect weekly visits during the first two months and less frequent visits (biweekly or monthly) for the last two months. Some sessions that are provided via telehealth might be video recorded and later reviewed to ensure that the program is being delivered as intended.
  Arms: Behavioral Care Coordinated with Medical Care
Behavioral: Behavioral Care Not Coordinated with Medical Care Intervention — Participants will meet with a study team member during their in-person visit and will receive a list of clinics that are panelled with their insurance. The participants will be responsible for calling the clinics to set up their appointments. Services might be provided in person or via telehealth based on the participant's preference and the clinics' availability.
  Arms: Behavioral Care Not Coordinated with Medical Care

SUMMARY:
The purpose of this study is to understand how behavioral health care that is coordinated with diabetes medical care compared with behavioral care that is provided in the community (and therefore not coordinated with diabetes medical care).

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 Diabetes diagnosed for one year or more
2. Latino or Black ethnicity/race
3. Speak and read English or Spanish
4. Eligibility for Medicaid

Exclusion Criteria:

1. Significant developmental disability
2. Serious psychiatric disorder
3. Another serious chronic illness

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic Control | Baseline and 4 months
  Will be measured by glycosylated hemoglobin A1c

SECONDARY OUTCOMES:
Change in Diabetes Self-Management | Baseline and 4 months
  We will measure Type 1 Diabetes Self-management using the Diabetes Management Questionnaire (DMQ; Score Range: 0-100, higher scores indicate greater adherence to diabetes management).

CONTACTS AND LOCATIONS:
Overall Officials: Luiza V Mali, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Univeristy of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No